CLINICAL TRIAL: NCT06442930
Title: EXtubation Related Complications - an International Observational Study To Understand the Impact and BEst Practices in the Operating Room and Intensive Care Unit - the EXTUBE Study
Brief Title: EXtubation Related Complications - the EXTUBE Study (EXTUBE)
Acronym: EXTUBE
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5811; 4850 (Other: Clinical Trials Ontario - CTO)
Record Dates: First submitted 2024-03-28; First posted 2024-06-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-07

CONDITIONS: Extubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EXTUBE is an international, multicentre, prospective cohort study evaluating the incidence, risk factors, and outcomes of extubation-related complications and describing clinical practices related to extubation after general anesthesia or after critical illness in the operating room (OR), out of OR anesthesia location or intensive care unit (ICU).

DETAILED DESCRIPTION:
Globally, over 200 million people each year require extubation. While routinely performed, extubation is a skilled and potentially high-risk procedure that should be performed only when physiologic, pharmacologic, and contextual conditions are optimal. Complications at this stage of patient care can result in decreased oxygen delivery to the brain and body, sometimes leading to serious adverse events such as cardiac arrest, brain damage, or death. Indeed, one quarter of airway complications that result in death or brain death occur at the time of extubation.

Despite the frequency of extubation and the potential for life-threatening complications, there is a lack of systematic data on the rate and circumstances under which these severe complications occur. The limited data indicate 10-30% of extubations may lead to severe complications, depending on the population and outcome definition. However, the certainty of these estimates is severely limited because they are based on studies that are small, mostly single-center, based on clinician recall, only capture a small portion of extubation complications (e.g., malpractice claims), or do not reflect current clinical practice. In addition, most lack a denominator and exclude successful extubations, making estimates of actual complication rates and risk factors impossible.

There has been no large study of extubation techniques or adherence to guidelines, so procedural factors associated with complications must be elucidated. While adherence to clinical practice guidelines has not been formally evaluated, surveys show non-adherence to some best practices and considerable variation in practice, and data from audits and medicolegal claims show that lack of adherence to best practices is frequently at the root cause of severe adverse extubation outcomes, with half of the complications deemed preventable. Therefore, data on the frequency and nature of extubation complications, patient and procedural risk factors for complications, and guideline adherence rates are needed before these preventable events can be addressed.

EXTUBE (EXtubation related complications - an international observational study To Understand the impact and BEst practices in the operating room and intensive care unit) is an international, multicenter, prospective cohort study

The primary objective of this study is to determine the incidence of severe extubation-related complications within 60 minutes after extubation in adults who have undergone mechanical ventilation for general anesthesia or critical illness. The secondary objectives are to determine: 1) the incidence of mild extubation complications; 2) patient- and procedure-related risk factors for extubation complications; 3) the association between extubation complications and outcomes until hospital discharge; and 4) the rate of adherence to extubation clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Undergoing extubation of an endotracheal tube (including index extubation and re-extubations) after general anesthesia in the OR, out of OR anesthesia location or ICU
* Undergoing extubation during the specified enrollment window

Exclusion Criteria:

* Patients will be excluded if the extubation is performed in the context of withdrawal of life support measures,
* Patients will be excluded if the extubation is performed for tracheostomy decannulation

For each patient who is not included, reasons for exclusion will be reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years old) undergoing extubation of an endotracheal tube (including index extubation and re-extubations) after general anesthesia in the OR, out of OR anesthesia location or ICU during the specified enrollment window
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
At least one of the following, occurring within 60minutes after extubation (composite outcome): i) Severe hypoxemia ii) Cardiac arrest iii) Need for airway management | Within 60 minutes after the end of extubation
  The primary outcome will be the occurrence of at least one of the following (composite outcome) occurring within 60 minutes after the end of extubation:
  i) Severe hypoxemia (oxygen saturation as measured by pulse oximetry falls below SpO2 < 80% for > 5 minutes) ii) Cardiac arrest iii) Need for airway management (reintubation, insertion of a supraglottic airway, bag-mask ventilation).

SECONDARY OUTCOMES:
Difficult airway and complications related to airway management if reintubation is required | Within 60 minutes after the end of extubation
  Difficult airway (i.e., experienced difficulty by an experienced airway manager with any or all of laryngoscopy or tracheal intubation, supraglottic airway use, face-mask ventilation, or front-of-neck airway) and complications related to airway management (e.g., esophageal intubation) if reintubation is required
Planned and unplanned non-invasive respiratory support | Within 60 minutes after the end of extubation
  Planned and unplanned non-invasive respiratory support or high flow nasal cannula
Emergency front of neck airway | Within 60 minutes after the end of extubation
  Emergency front of neck airway should airway management be required after extubation
Cardiac arrhythmia requiring chemical or electrical treatment | Within 60 minutes after the end of extubation
  Cardiac arrhythmia requiring chemical or electrical treatment
Severe Hypotension | Within 60 minutes after the end of extubation
  Severe hypotension (systolic arterial pressure < 65 mmHg recorded at any time or systolic arterial pressure < 90 mmHg for > 30 minutes or new need/increase of vasopressor and/or fluid load > 15 mL/kg)
Severe Hypertension | Within 60 minutes after the end of extubation
  Severe hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥120 mmHg),
Pulmonary aspiration | Within 60 minutes after the end of extubation
  Aspiration of gastric contents (gastric contents inhaled into the larynx and the respiratory tract)
Barotrauma | Within 60 minutes after the end of extubation
  Pneumothorax/pneumo-mediastinum
Dental injury | Within 60 minutes after the end of extubation
  Dental injury (notable change to the patient's dentition attributable to extubation or to reintubation, should this be required)
Airways injury | Within 60 minutes after the end of extubation
  Airways injury (e.g., vocal cord damage, arytenoid dislocation
Mortality | Within 7 days after extubation
  In-hospital mortality
Re-intubation | Within 48 hours after extubation
  Re-intubation within 48 hours of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Parotto, MD, PhD, Principal Investigator — UHN
Locations (21):
- United States (5):
  - Banner University Medical Centre, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Florida, Gainesville, Florida
  - Oregon Health & Science University, Portland, Oregon
  - The University of Texas Health Science Center, Houston, Texas
- Australia (5):
  - Royal North Shore Hospital, Sydney, New South Wales
  - The Northern Hospital, Melbourne, Victoria
  - Eastern Health - Box Hill Hospital, Melbourne, Victoria
  - Eastern Health - Maroondah Hospital, Melbourne, Victoria
  - Eastern Health - Angliss Hospital, Melbourne, Victoria
- Canada (7):
  - Surrey Memorial Hospital, Surrey, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Niagara Health - Marotta Family Hospital, Saint Catharines, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
- Galway University Hospitals, Galway, Ireland
- Tan Tock Seng Hospital, Singapore, Singapore
- United Kingdom (2):
  - Royal United Hospitals Bath, Bath
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No